CLINICAL TRIAL: NCT07027228
Title: Effect of Using Virtual Reality Glasses and Music During Blood Donation on Anxiety, Vital Signs and Satisfaction of Donors: A Randomized Controlled Trial
Brief Title: Virtual Reality Glasses and Music During Blood Donation on Anxiety, Vital Signs and Satisfaction of Donors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Yadigar Ordu, PhD, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Distraction Techniques
Record Dates: First submitted 2025-05-26; First posted 2025-06-18 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Satisfaction
Keywords: blood donation; virtual reality; music; anxiety; vital signs; donor satisfaction
MeSH Terms: conditions — Personal Satisfaction; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual reality glasses group (Experimental): This is the group where anxiety, vital signs and donor satisfaction will be evaluated using virtual reality glasses.
  Interventions: Other: Using virtual reality glasses or listening to music
- Music group (Experimental): This is the group where anxiety, vital signs and donor satisfaction will be evaluated using a music application.
  Interventions: Other: Using listening to music
- Control group (No Intervention): This is the group where anxiety, vital signs and donor satisfaction will be evaluated without any intervention.

INTERVENTIONS:
Other: Using virtual reality glasses or listening to music — Donors in the intervention group will be randomly assigned and shown relaxing nature images through virtual reality glasses.
  Arms: Virtual reality glasses group
Other: Using listening to music — Donors in the intervention group will be randomly assigned and will listen to relaxing music.
  Arms: Music group

SUMMARY:
Blood is considered a limited resource in health centers and blood and blood products must be kept ready. The COVID-19 pandemic has caused a significant decrease in life-saving blood donations. In addition, negative experiences such as vasovagal reactions, painful needle sticks, psychological triggers and injuries that develop during blood donation cause donors to experience anxiety, negatively affecting their vital signs and the next donation experience. Therefore, donors should be supported by distraction techniques during blood donation.

DETAILED DESCRIPTION:
Among the techniques used to divert attention, virtual reality glasses and music applications are frequently used. It is reported that virtual reality glasses are effective in reducing anxiety and supporting vital signs and satisfaction positively because they make you feel like you are somewhere else and music has positive effects on the human soul. This study aims to determine the effect of using virtual reality glasses and music during blood donation on donors' anxiety, vital signs and satisfaction.

A single-blind randomized controlled clinical trial design with one control and two intervention groups will be used in the study. The universe of the study will consist of donors who applied to the Blood Center of Necmettin Erbakan University Faculty of Medicine Hospital between June and July 2025. The sample of the study will consist of 225 male donors who meet the inclusion criteria and agree to participate in the study. Donors will be randomly assigned to 75 Intervention-1 Group (virtual reality glasses), 75 Intervention-2 Group (music) and 75 control groups using the simple randomization method. Data will be collected through face-to-face interviews with donors using the "Descriptive Characteristics Form", "State and Trait Anxiety Scale", "Vital Findings Follow-up Form" and "Satisfaction Scale". The first researcher will act as the evaluator and the second researcher will act as the implementer in the collection of data. Thus, differences between the evaluator and the implementer will be eliminated. Donors will be shown images of nature using virtual reality glasses, donors in the other group will listen to calming music, and the control group will not receive any intervention within the scope of standard practice. The data obtained from the study will be analyzed using the SPSS 22 package program and the data will be evaluated at a 95% confidence interval and a significance level of 0.05.

ELIGIBILITY:
Inclusion Criteria:

The criteria for inclusion in the study are as follows:

* Being between the ages of 18-60,
* Having a visual, hearing or perception disorder that prevents communication,
* Having neurological, psychiatric or psychological diseases,
* Donating whole blood.

Exclusion Criteria:

The exclusion criteria for the study are as follows:

* Having vasovagal reactions,
* Having complaints such as migraine, vertigo, active nausea, vomiting, headache,
* Not having the blood donation chair in the semi-fowler position throughout the application,
* Wanting to leave the study.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 225 (Actual)
Dates: Start 2025-06-23 (Actual); Primary Completion 2025-07-10 (Actual); Study Completion 2025-07-23 (Actual)

PRIMARY OUTCOMES:
State and Trait Anxiety Scale | Up to two months
  The State and Trait Anxiety Scale is one of the scales frequently used in measuring anxiety. The scale consists of two parts: a 20-item "state anxiety form" and a 20-item "trait anxiety form". Individuals are asked to answer four-point Likert items (1: not at all, 2: a little, 3: a lot of the time, 4: completely) to determine what they are feeling at that moment. Since this study aims to measure donors' anxiety levels before and after blood donation, the state anxiety measuring part of the scale will be used. The scores obtained from the scale vary between 20 and 80. Although there is no anxiety threshold on the scale, a high score indicates a high anxiety level, and a low score indicates a low anxiety level.
Blood pressure | Up to two months
  Individuals' blood pressure values will be determined with a sphygmomanometer.
Pulse | Up to two months
  Individuals' pulse values will be determined by measuring with a pulse oximeter.
Oxygen saturation | Up to two months
  Individuals' oxygen levels will be determined by measuring with a pulse oximeter.
Respiratory | Up to two months
  The ventilation value of the individuals will be measured and recorded from the anterior thorax for one minute.
Satisfaction Scale | Up to two months
  It is an evaluation form consisting of five statements (5: Very satisfied, 4: Satisfied, 3: Undecided, 2: Not satisfied, 1: Not satisfied at all) to determine donors' satisfaction with the virtual reality glasses and music application. An increase in the score indicates an increase in satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No